CLINICAL TRIAL: NCT02294552
Title: High-dose Post-transplantation Cyclophosphamide as Graft Versus-host Disease Prophylaxis After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Post-transplantation Cyclophosphamide as GVHD Prophylaxis After HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ivan S Moiseev (Other)
Responsible Party: Sponsor-Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Organization: St. Petersburg State Pavlov Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCy-2014
Record Dates: First submitted 2014-10-30; First posted 2014-11-19 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Lymphoma; Myelodysplastic Syndromes; Chronic Lymphocytic Leukemia; Immune System Diseases
Keywords: Cyclophosphamide; Leukemia; Lymphoma; Myelodysplastic Syndromes; Chronic Lymphocytic Leukemia; Immunosuppressive Agents; Immune System Diseases; Busulfan; Fludarabine; Tacrolimus; Mycophenolate mofetil; Antineoplastic Agents, Alkylating; Myeloablative Agonists; Hematopoietic Stem Cell Transplantation; Allogeneic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Immune System Diseases; Leukemia | interventions — Cyclophosphamide; Busulfan; fludarabine phosphate; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matched bone marrow graft (Experimental): Days -8 through -4: Busulfan 1 mg/kg po qid x 4 days Days -3 through -2: Cyclophosphamide 50mg/kg/day iv x 2 days Or Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -4 through -3: Busulfan 1 mg/kg po qid x 2 days Day 0: Infusion of unmanipulated graft Day +3 and +4: Cyclophosphamide 50 mg/kg/day iv
  Interventions: Drug: Cyclophosphamide; Drug: Busulfan; Drug: Fludarabine monophosphate; Procedure: Allogeneic hematopoietic stem cell transplantation
- Matched peripheral blood stem cells graft (Experimental): Days -8 through -4: Busulfan 1 mg/kg po qid x 4 days Days -3 through -2: Cyclophosphamide 50mg/kg/day iv x 2 days Or Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -4 through -3: Busulfan 1 mg/kg po qid x 2 days Day 0: Infusion of unmanipulated graft Day +3 and +4: Cyclophosphamide 50 mg/kg/day iv Days +5 through +35: Mycophenolate mofetil 30 mg/kg/day, maximum 2 g/day, iv or po x 30 days Days +5 through +120: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Cyclophosphamide; Drug: Busulfan; Drug: Fludarabine monophosphate; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Procedure: Allogeneic hematopoietic stem cell transplantation
- Mismatched peripheral blood stem cells or bone marrow graft (Experimental): Days -8 through -4: Busulfan 1 mg/kg po qid x 4 days Days -3 through -2: Cyclophosphamide 50mg/kg/day iv x 2 days Or Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -4 through -3: Busulfan 1 mg/kg po qid x 2 days Day 0: Infusion of unmanipulated graft Day +3 and +4: Cyclophosphamide 50 mg/kg/day iv Days +5 through +35: Mycophenolate mofetil 45 mg/kg/day, maximum 3 g/day, iv or po x 30 days Days +5 through +120: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Cyclophosphamide; Drug: Busulfan; Drug: Fludarabine monophosphate; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Procedure: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Busulfan
Drug: Fludarabine monophosphate
Drug: Tacrolimus
  Arms: Matched peripheral blood stem cells graft; Mismatched peripheral blood stem cells or bone marrow graft
Drug: Mycophenolate mofetil
  Arms: Matched peripheral blood stem cells graft; Mismatched peripheral blood stem cells or bone marrow graft
Procedure: Allogeneic hematopoietic stem cell transplantation

SUMMARY:
This study evaluates the efficacy of high-dose post-transplantation cyclophosphomide as graft-versus-host disease (GVHD) prophylaxis after allogeneic stem cell transplantation in patients with different risk of GVHD. The risk-adapted strategy involves using single-agent cyclophosphomide in recipients of matched bone marrow graft, and combining cyclophosphomide with tacrolimus and mycophenolate mofetil in recipients of matched peripheral blood stem cells and mismatched bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an indication for allogeneic hematopoietic stem cell transplantation
* Signed informed consent
* Patients with a donor available. The donor and recipient must be identical at at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum match of 5/10 is required for related donor. A minimum match of 8/10 is required for unrelated donor.
* No second tumors
* No severe concurrent illness

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidence of acute and chronic GVHD, requiring treatment | 365 days

SECONDARY OUTCOMES:
Incidence of primary graft failure | 60 days
Non-relapse mortality analysis | 365 days
Overall survival analysis | 365 days
Event-free survival analysis | 365 days
Relapse rate analysis | 365 days
Toxicity based NCI CTC grades | 100 days
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Boris V Afanasyev, MD, Prof., Principal Investigator — First Pavlov State Medical University of St. Petersburg
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

REFERENCES:
- [Derived] Moiseev IS, Pirogova OV, Alyanski AL, Babenko EV, Gindina TL, Darskaya EI, Slesarchuk OA, Bykova TA, Chukhlovin AB, Pevtcov DE, Bondarenko SN, Afanasyev BV. Risk-adapted GVHD prophylaxis with post-transplantation cyclophosphamide in adults after related, unrelated, and haploidentical transplantations. Eur J Haematol. 2018 May;100(5):395-402. doi: 10.1111/ejh.13030. Epub 2018 Mar 1. PMID 29360184